CLINICAL TRIAL: NCT05887232
Title: Comparative Study on the Efficacy of Fractional CO2 and Fractional CO2 Laser With Autologous Platelet Rich Plasma in Scars
Brief Title: Comparison of Co2 Laser Versus Co2 Laser With PRP in Scars
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, Zahra Nigar, Principle Investigator, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMHAbbottabad1988
Record Dates: First submitted 2023-05-16; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: CO2 Laser in Scars

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fractional Co2 laser (Active Comparator): Patient in group A received FCL treatment's four sessions four weeks apart.
  Interventions: Procedure: Fractional CO2 laser
- Platelet Rich Plasma (Active Comparator): Group B received fractional CO2 with four Platelet Rich Plasma sessions,4 weeks apart.
  Interventions: Procedure: Fractional CO2 with Platelet Rich Plasma

INTERVENTIONS:
Procedure: Fractional CO2 laser — Patient in group A received FCL treatments four sessions with four weeks apart
  Arms: Fractional Co2 laser
Procedure: Fractional CO2 with Platelet Rich Plasma — Group B received four PRP and FCL sessions 4 weeks apart
  Arms: Platelet Rich Plasma

SUMMARY:
Objective: To compare the effect of Fractional Carbon dioxide Laser (FCL) Vs Fractional Carbon dioxide Laser with platelet rich plasma (PRP) in management of Scars.

Study design: Randomized-controlled trial (RCT). Study setting and duration: Dermatology Department, CMH-Abbottabad, November 2022/April 2023.

Methodology: The sample size of 60 patients, age 18 to 50 years, was calculated by using Openepi app and the non-probability consecutive sampling technique was used. Patient in group A received FCL treatment's four sessions with four weeks apart, whereas Group B received four PRP and FCL sessions. The Quartile grading scale (score 0 is <25%, score 1 is 25-50%, score 2 is 51-75% and score 3 is >75% improvement) was used to assess the patient's clinical improvement at 4 weeks after each session. To determine statistical significance χ2-square test, taking p-value <0.05 as significant, was used.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-50 years
* Fitzpatrick skin type III-V
* Presented with post-acne, post traumatic or post burn scars
* all those patients emotionally balanced with realistic expectations were included in the study.

Exclusion Criteria:

* scar that was less than 6 months old
* if they had an active infection or inflammatory skin condition
* having a history of malignancy
* a known connective tissue illness
* history of excessive bleeding or keloids
* unrealistic expectations
* pregnant or breastfeeding.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Quartile grading scale for assessment of scars | 16 weeks
  Quartile grading scale was used to assess effectiveness of CO2 laser and CO2 laser with Platelet rich plasma in scars.Minimum score=0,Maximum Score=3 .Maximum score means better outcome.The Quartile grading scale (score 0 is <25%, score 1 is 25-50%, score 2 is 51-75% and score 3 is >75% improvement) was used to assess the patient's clinical improvement at 4 weeks after each session.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr.Zahra Nigar, Abbottabad, KPK, Pakistan